CLINICAL TRIAL: NCT01354509
Title: Normothermia Protocol for Traumatic Brain Injury Patients: An Outcome Study
Brief Title: Normothermia Protocol for Traumatic Brain Injury Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medivance, Inc. (Industry)
Responsible Party: Farid Sadaka, MD, Mercy St John's Medical Center
Other Study IDs: MDV_STL_001
Record Dates: First submitted 2011-05-12; First posted 2011-05-17 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2011-05

CONDITIONS: Traumatic Brain Injury
Keywords: Normothermia; fever control; Outcome study
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Current protocol group: Patients treated with current standards based on physician discretion.
- Normothermia group: Normothermia protocol, using Hydrogel cooling Pads(Arctic Sun) applied for 96 hrs starting upon admission to the ICU

SUMMARY:
Comparison between a normothermia protocol and current protocol (acetaminophen plus blankets)

1. Normothermia Protocol is successful in achieving and maintaining normal temperature in moderate to severe Traumatic Brain Injury (TBI) patients.(using Arctic Sun for 96 hrs from admission to Neuro ICU)
2. Normothermia is translated into improved neurologic Outcome and survival compared to standard of care (Physician management)

ELIGIBILITY:
Inclusion Criteria:

* Severe TBI patients(GCS 3-9) admitted to ICU

Exclusion Criteria:

* Less than 18 years OLD.
* Bleeding disorders.
* Pregnancy/Breastfeeding.
* Hepatic Encephalopathy.
* Spinal cord injury (know or new)
* Fever >100 F prior to randomization.
* Blood Alcohol level >80
* Participation in other Research trial.
* Inability/unwilling to obtain Informed consent.
* Terminal illness(not expected to survive 3-6 months)
* Not expected to survive 24 hrs.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe TBI patients(GCS 3-9) admitted to ICU
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the Normothermia protocol | 5 days
  Number of times patient's temp was above 37°C during this 96 hr period
Temperature vs ICP | 5 days
  Number of times ICP > 20 in patients with ICP monitors
Neurologic Outcome of the 2 patient populations | 1month, 3 months, 6 months
  Modified Rankin Scale at Hospital discharge, 3 months, and 6 months

SECONDARY OUTCOMES:
Mortality | 5 days, 3 months, 6 months
  In-Hospital mortality, 3 - 6 month mortality

CONTACTS AND LOCATIONS:
Overall Officials: Farid Sadaka, MD, Principal Investigator — Mercy St John's Medical Center
Locations (1):
- Mercy St John's Medical Center, St Louis, Missouri, United States